CLINICAL TRIAL: NCT03580577
Title: Risk Factors and Outcomes of Acute Venous Thromboembolism in Cirrhotic Patients: A Hospital Based Prospective Study
Brief Title: Risk Factors and Outcomes of Acute Venous Thromboembolism in Cirrhotic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Radwan Riad, Assistant lecturer, Assiut University
Other Study IDs: Liver cirrhosis and thrombosis
Record Dates: First submitted 2018-06-16; First posted 2018-07-09 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Liver Cirrhosis; Venous Thromboembolism
MeSH Terms: conditions — Liver Cirrhosis; Venous Thromboembolism | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhotic with venous thromboembolism: cirrhotic patients with a venous thromboembolic event (including deep venous thrombosis, pulmonary embolism, acute non-malignant portal vein thrombosis, splenic vein, inferior vena cava thrombosis or mesenteric vascular occlusion).
  Each patient will subjected to through history taking and careful examination to detect and risk factors also laboratory work to detect thrombocytopenia, disease severity, coagulation status thrombelastography before starting anticoagulants.
  * Patients will start treatment with anticoagulants therapy after liaise with the specialized physician.
  * Protein C, protein S and antithrombin III level will be assessed 3 months after the acute thrombotic event and 1 month of vitamin K antagonist (VKA) withdrawal.
  Interventions: Device: thromboelastography
- Cirrhotic without venous thromboembolism: cirrhotic patients without any thrombotic events Each patient will subjected to through history taking and careful examination to detect and risk factors.
  - Protein C, protein S and antithrombin III level will be assessed at baseline.

INTERVENTIONS:
Device: thromboelastography — thromboelastography will assess all coagulation abnormalities including platelets function in cirrhotic group with venous thromboembolism , and guide us about is there increased thrombosis risk or not, for that a fresh blood sample will be withdrawn from each patient before starting any treatment
  Groups: Cirrhotic with venous thromboembolism

SUMMARY:
patient with liver cirrhosis was supposed to have autoanticoagulation which approved to be wrong, with absence of conventional method to detect all abnormalities in coagulation state. Thromboelastography (TEG) give a broad picture for the coagulation defects.

In addition to that no guidelines prescribed anticoagulants for venous thromboembolism in cirrhotic, so the investigators will do a study to demonstrate frequency and risk factors for acute venous thromboembolism in cirrhotic patients, find a conventional laboratory method and test TEG to assess risk of thrombosis in cirrhotic patients.Also, to validate current algorithm for use of anticoagulant and antiplatelet for thromboembolism for non cirrhotic in cirrhotic patients.

DETAILED DESCRIPTION:
Nowadays, the term "autoanticoagulated" ,which prescribed coagulopathy state in chronic liver disease (CLD) patients due to impaired synthesis of coagulation factors and elevated international normalized ratio(INR), has been approved to be wrong and those patients are liable for venous thromboembolism (VTE) with 0.5% - 6.3% incidence of deep venous thrombosis (DVT) and pulmonary thromboembolism (PE) among cirrhotic patients.

This may be explained by normal or even increased production of factor VIII and von Willebrand factor, enhanced thrombin activity and Low level of protein C, protein S and antithrombin III due to impaired liver synthesis, other risk factor include sedentary lifestyle, fractures, immobility, hospitalization, elevated estrogen levels, surgery, concomitant disease states and cancer, damaged vasculature that increases inflammation, and sluggish splanchnic blood flow, which are all common in those patients.

Absence of gold standard estimation for hypercoagulability in cirrhotic patients, is a big problem. During measurement of conventional parameters such as international normalized ratio (INR) or partial thromboplastin time, reagents used to measure the prothrombin time do not contain thrombomodulin on which protein C depend for activation, so it does not adequately reflect reduced levels protein C. Thromboelastography a device that has the ability to measure whole blood coagulation cascade including platelet function, It can be used to monitor coagulation status before liver transplantation operation to properly identify and treat coagulation abnormalities.

No worldwide guidelines is established neither for management nor prophylaxis of VTE in cirrhotic patients, this may be due to safety concerns regarding the risk of bleeding related to anticoagulant drugs when used in people with advanced liver disease, especially if there is significant thrombocytopenia, and/or the presence of varices.

ELIGIBILITY:
Inclusion Criteria:

* all cirrhotic patient who developed venous thromboembolic events
* written informed consent (patient or nearest relative )

Exclusion Criteria:

* Patient with chronic thromboembolic event ( e.g. chronic pulmonary embolism, chronic portal vein thrombosis).
* patients on antiplatelets or anticoagulants.
* Patients with end stage kidney, heart or lung diseases
* Pregnant.
* Cirrhotic patients on control group who develop an acute thromboembolic event during the study period will be excluded and shifted to the case group

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: liver cirrhosis patients with acute venous thromboembolism (VTE), control group of cirrhotic patients without VTE
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Occurence of recanalization of thrombosed vessel | 24 weeks from baseline
  Efficacy of anticoagulants describe its ability to prevent further thrombosis and restore patency of thrmobosed vessel

SECONDARY OUTCOMES:
detect safety of anticoagulants in cirrhotic | During treatment period wither 12 or 24 weeks from starting therapy
  Occurrence of any bleeding event while on anticoagulants therapy
Correlate thromboelastography results with hypercoagluable state in cirrhotic patients with venous thromboembolism | 1 day
  Changes in r, k and MA- TEG parameters in cirrhotic patients with venous thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel Sabour Mohamed Mekky, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Gulley D, Teal E, Suvannasankha A, Chalasani N, Liangpunsakul S. Deep vein thrombosis and pulmonary embolism in cirrhosis patients. Dig Dis Sci. 2008 Nov;53(11):3012-7. doi: 10.1007/s10620-008-0265-3. Epub 2008 Apr 29. PMID 18443906
- [Background] Northup PG, McMahon MM, Ruhl AP, Altschuler SE, Volk-Bednarz A, Caldwell SH, Berg CL. Coagulopathy does not fully protect hospitalized cirrhosis patients from peripheral venous thromboembolism. Am J Gastroenterol. 2006 Jul;101(7):1524-8; quiz 1680. doi: 10.1111/j.1572-0241.2006.00588.x. PMID 16863556
- [Background] Dhar A, Mullish BH, Thursz MR. Anticoagulation in chronic liver disease. J Hepatol. 2017 Jun;66(6):1313-1326. doi: 10.1016/j.jhep.2017.01.006. Epub 2017 Jan 12. PMID 28088580
- [Background] Tripodi A, Primignani M, Chantarangkul V, Dell'Era A, Clerici M, de Franchis R, Colombo M, Mannucci PM. An imbalance of pro- vs anti-coagulation factors in plasma from patients with cirrhosis. Gastroenterology. 2009 Dec;137(6):2105-11. doi: 10.1053/j.gastro.2009.08.045. Epub 2009 Aug 23. PMID 19706293
- [Background] Tripodi A, Primignani M, Lemma L, Chantarangkul V, Mannucci PM. Evidence that low protein C contributes to the procoagulant imbalance in cirrhosis. J Hepatol. 2013 Aug;59(2):265-70. doi: 10.1016/j.jhep.2013.03.036. Epub 2013 Apr 11. PMID 23583273
- [Background] Tripodi A, Primignani M, Chantarangkul V, Clerici M, Dell'Era A, Fabris F, Salerno F, Mannucci PM. Thrombin generation in patients with cirrhosis: the role of platelets. Hepatology. 2006 Aug;44(2):440-5. doi: 10.1002/hep.21266. PMID 16871542
- [Background] Tripodi A, Salerno F, Chantarangkul V, Clerici M, Cazzaniga M, Primignani M, Mannuccio Mannucci P. Evidence of normal thrombin generation in cirrhosis despite abnormal conventional coagulation tests. Hepatology. 2005 Mar;41(3):553-8. doi: 10.1002/hep.20569. PMID 15726661
- [Background] van Wijngaarden A, van den Besselaar AM, Bertina RM. Thrombomodulin activity in commercial thromboplastin preparations. Thromb Res. 1986 Aug 1;43(3):265-74. doi: 10.1016/0049-3848(86)90146-5. PMID 3016943
- [Background] Tripodi A, Primignani M, Braham S, Chantarangkul V, Clerici M, Moia M, Peyvandi F. Coagulation parameters in patients with cirrhosis and portal vein thrombosis treated sequentially with low molecular weight heparin and vitamin K antagonists. Dig Liver Dis. 2016 Oct;48(10):1208-13. doi: 10.1016/j.dld.2016.06.027. Epub 2016 Jul 1. PMID 27470055
- [Background] HARTERT H. [Thrombelastography, a method for physical analysis of blood coagulation]. Z Gesamte Exp Med. 1951;117(2):189-203. No abstract available. Undetermined Language. PMID 14836887
- [Background] Collins S, MacIntyre C, Hewer I. Thromboelastography: Clinical Application, Interpretation, and Transfusion Management. AANA J. 2016 Apr;84(2):129-34. PMID 27311154
- [Background] MacIvor D, Rebel A, Hassan ZU. How do we integrate thromboelastography with perioperative transfusion management? Transfusion. 2013 Jul;53(7):1386-92. doi: 10.1111/j.1537-2995.2012.03728.x. Epub 2012 Jun 7. No abstract available. PMID 22670837